CLINICAL TRIAL: NCT03261713
Title: Home-based Virtual Reality Training After Discharge From Hospital-based Stroke Rehabilitation: A Parallel Randomised Feasibility Trial.
Brief Title: Home-based Virtual Reality Training After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: Bruyere Academic Medical Organization (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAMO IF2017
Record Dates: First submitted 2017-06-13; First posted 2017-08-25 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Stroke
Keywords: rehabilitation; telerehabilitation; feasibility studies; virtual reality
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A prospective, single-site, single-blinded, parallel-group (1:1 ratio) randomized feasibility trial on the use of VRT for ongoing stroke rehabilitation after discharge from inpatient or outpatient stroke rehabilitation.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor does not know the participant's intervention group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Virtual reality training designed to train standing balance, reaching, stepping, gentle strengthening and aerobic conditioning.
  Interventions: Device: Virtual reality
- Control (Active Comparator): iPad apps designed to train memory, cognition, visual tracking and fine motor skills.
  Interventions: Device: Control

INTERVENTIONS:
Device: Virtual reality — Virtual reality training is provided using Jintronix Rehabilitation software. A Kinect camera captures the movements of the participant using infrared technology and allows them to control an avatar, which interacts with an activity. Several games and activities are available to train standing balance (ex. slalom skiing), reaching (ex. planting seeds/harvesting tomatoes), stepping (ex. whack-a-mole), gentle strengthening (ex. knee extensions) and aerobic exercises (ex. marching on the spot). Game and activity difficulty can be increased by requiring more repetitions, or greater speed, distance and/or accuracy. Specific games and activities, and their parameters are customized for each participant. The exercise plan is performed 5 times a week for 6 weeks for 30 minutes at each session.
  Arms: Virtual Reality
Device: Control — Participants in the control group are provided with an iPad which contains a selection of apps suited for memory (ex. memory card game), cognition (Sudoku, cross-word), visual tracking (word search) and fine motor skills (ex. writing, whack-a-mole). Participants are instructed to perform their exercise plan 5 times a week for 6 weeks for 30 minutes at each session.
  Arms: Control

SUMMARY:
Virtual reality (VR) training (VRT) uses computer software to track a user's movements and allow them to interact with a game presented on a TV. It is fun and engaging and may encourage the user to do more exercise. VRT is increasingly being used for rehabilitation after stroke. Patients often require ongoing therapy post-discharge from inpatient rehabilitation. Outpatient therapy may be unavailable due to waiting lists, transportation issues, distance etc.; therefore, home-based VRT may be the answer. Our objectives are to determine: 1) the feasibility of home-based VRT for stroke patients after discharge from hospital-based rehabilitation, and 2) the feasibility of a battery of outcome measures. Forty stroke rehabilitation patients will be recruited over 18 months and randomize them to experimental or control groups. VRT participants will be introduced to VRT at the hospital and a VRT system will be set up in their homes shortly after discharge. Control participants will be provided with games and apps on an iPad focusing on cognition and fine motor skills. Participants will be instructed to perform 30 minutes of VRT 5 days a week for 6 weeks. Training will be monitored remotely. Both groups will receive weekly phone calls to review their home activity and answer questions. Measurements will be made of standing balance and general function before and after training, and feasibility (compliance, enjoyment, safety).

DETAILED DESCRIPTION:
Stroke causes approximately 15 300 hospital admissions per year in Ontario and 50% of individuals who have had a stroke are left with moderate to severe impairment. Because of the severity of their condition, these individuals often cannot stand and have poor sitting and standing balance. Most patients who are discharged from inpatient stroke rehabilitation are 8-10 weeks post-stroke and have not completely recovered. Their brains are still in a period of enhanced neuroplasticity, during which great functional change can be made; Therapy outcomes are dose-dependent; intensive, high-repetition, task-oriented and task-specific therapies are most effective. Therefore, for the greatest recovery possible, these patients require ongoing therapy. Most are offered this on an outpatient basis. However, for many reasons (transportation difficulties, distance from downtown, weather etc.), not all eligible patients are able to attend outpatient therapy. Also, there is a waiting list and a limited number of outpatient therapy sessions are offered to each patient.

Virtual reality training (VRT) uses computer software to track the user's movements and allow him or her to interact with a game or activity presented on a TV screen. It is convenient, timely, and enjoyable, and may be done for an unlimited period post-stroke. VRT has been shown to benefit upper extremity function, standing balance, gait and overall function. Home-based VRT offers a promising addition or alternative to existing rehabilitation programs and home exercise programs that could make a significant difference in the lives of stroke survivors. A few pilot studies have investigated the use of home-based VRT for standing balance and upper extremity recovery after stroke and shown the feasibility of these systems for ongoing rehabilitation in the home. The investigators wish to expand on these studies by using a new VR system, made by Jintronix Inc. (Montreal, QC). This system was initially developed for stroke rehabilitation and has also been used extensively with healthy and frail elderly individuals. The Jintronix system is marketed for institutional and home use and has a simple-to-use interface but its home use has not yet been fully evaluated. The games are designed to incorporate motor learning principles such as multiple forms of feedback and task-specific practice that can be progressed to maintain an appropriate level of challenge. The purpose of this study is to investigate the feasibility, acceptance and safety of this new, simple-to-use VRT system used in the home, combined with substantial remote support for the user.

The primary objectives assessed the feasibility of using VRT in the home by patients post-stroke, using quantitative and qualitative methods. Specific objectives were:

1. To estimate the recruitment rate of participants into the study;
2. To assess the ability and compliance of the participants with respect to the components of the research protocol (ability to learn VRT through the training program; ability to comply with the exercise protocol; participant retention);
3. To determine the safety of home-based VRT (presence of minor and major adverse events);
4. To assess the ability of stroke survivors and their study partners to use VRT technology in the home (i.e. technical difficulties, difficulty learning the games);
5. To assess the acceptability of the VRT intervention (enjoyment; perceived efficacy)
6. To estimate the cost for a future definitive randomised control trial (RCT) on in-home VRT.

The secondary objectives assessed the feasibility of the outcome measures, using quantitative and qualitative methods. Specific objectives were:

1. To assess the feasibility and acceptance of a battery of outcome measures, including physical assessments, questionnaires, an interview and a log book;
2. To assess the potential that home-based VRT might maintain or improve physical outcomes (standing balance, gait, general function) and community integration after discharge from hospital-based stroke rehabilitation, compared to those who only participate in their regular activities of daily living.
3. To determine the sample size required for a future definitive RCT on in-home VRT.

Procedures Participants in both the experimental and control groups (and their caregivers for those in the experimental group only) attend a total of 4 sessions at Élisabeth Bruyère Hospital. The first three sessions occur in the week or two before discharge from inpatient or outpatient rehabilitation. At sessions 1 and 2, each lasting approximately 60 minutes, participants and their study partners in the experimental group are trained on how to use the VRT system and play the games. They are also instructed what to do if something went wrong (for example, if the participant falls or the equipment does not work). Participants are given a simple manual on VRT. Participants in the control group also attend two training sessions, each lasting approximately 45 minutes, on how to use the tablet and use the apps. Outcome measures are performed at sessions 3 (before discharge) and 4 (after 6 weeks of VRT); each session takes approximately 1½ hours.

After discharge from inpatient or outpatient rehabilitation, the research physical therapist (PT) installs the VRT system into the participant's home and reviews the games, safety considerations and follow-up procedures with the participant and their study partner. The supervising caregiver must be in the home of the participant while he or she is doing VRT. The PT monitors the game and parameter selections along with time spent on VRT at least once a week using the remote access feature of the VRT system, and modifies the games if necessary.

Participants in both groups are instructed to perform their exercise plan 5 times a week for 6 weeks for 30 minutes at each session. This amount of additional training (15 hours) has been shown to produce a significant improvement in activities of daily living post-stroke. All participants are contacted by telephone twice a week for the first week and at least once a week for the following 5 weeks to offer encouragement, suggest modifications to the games and identify any safety issues or technical problems. Participants are also invited to contact the research PT as needed. Participants in both groups are encouraged to do as many activities of daily living (ADLs) and instrumental ADLs (IADLs) as they wish, including walking, participation in exercise groups and therapy. They are not prevented from undergoing further rehabilitation while enrolled in the feasibility study.

ELIGIBILITY:
Inclusion Criteria:

1. have had a stroke (ischemic or hemorrhagic) resulting in physical impairment;
2. have enough preserved cognitive ability to learn VRT
3. are receiving inpatient or outpatient stroke rehabilitation services;
4. are able to stand independently for at least 2 minutes
5. have a study partner who could attend 2 training sessions with the participant and was able to be in the home with the participant while doing VRT;
6. can read, speak and understand English;
7. live within 50 km of Élisabeth Bruyère Hospital;
8. are able and willing to attend 4 appointments at Élisabeth Bruyère Hospital (2 for assessment; 2 for training);
9. will not be travelling away from home for more than 2 days a week for the duration of the study;
10. have enough space in their home to do VRT safely.

Exclusion Criteria:

1. have an unstable medical condition, seizures or vertigo,
2. are unable to perform mild to moderate exercise safely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 18 months
  number of participants recruited over 18 months of participant intake relative to the number who met study criteria and number who were approached
Quantitative assessment of ability and compliance to research protocol | 18 months
  assessed by monitoring the use and progression of the VRT program
Qualitative assessment of ability and compliance to research protocol | 18 months
  assessed through comments made by the participant and study partner
Adverse events (incidence & type) due to home-based VRT intervention | 18 months
  presence of adverse effects (minor and severe) recorded from telephone conversations and through log book
Ability to use VRT in the home | 18 months
  assessed through comments made by the participant and study partner
Quantitative assessment of acceptability of VRT intervention | 18 months
  assessed with the Physical Activity Enjoyment Scale
Qualitative assessment of acceptability of VRT intervention | 18 months
  assessed through comments made by the participant and study partner
Estimate cost for a future definitive RCT | 18 months
  calculate costs of all components of this study

SECONDARY OUTCOMES:
Ability of participants to perform Berg Balance Scale without quitting due to fatigue or frustration | 18 months
  1) Berg Balance Scale (BBS, Berg et al.)
Ability of participants to perform Timed Up & Go (original version) without quitting due to fatigue or frustration | 18 months
  Timed Up And Go (TUG, original version, Campbell et al.)
Ability of participants to perform Timed Up & Go (manual version) without quitting due to fatigue or frustration | 18 months
  Timed Up And Go (TUG, manual version, Hofheinz & Schusterschitz)
Ability of participants to perform Timed Up & Go (cognitive version) without quitting due to fatigue or frustration | 18 months
  Timed Up And Go (TUG, cognitive version, Lundin-Olsson et al.)
Ability of participants to perform Five Times Sit-to-Stand without quitting due to fatigue or frustration | 18 months
  Five Times Sit-to-Stand Test (FTSST, Bohannon et al.)
Ability of participants to perform Community Balance & Mobility Scale without quitting due to fatigue or frustration | 18 months
  Community Balance & Mobility Scale (CBM, Howe et al.)
Ability of participants to perform quantitative analysis of quiet stance in standing without quitting due to fatigue or frustration | 18 months
  movement of the centre of pressure on a force plate during quiet stance in standing (Preuss & Popovic)
Ability of participants to perform quantitative analysis of limits of stability in standing without quitting due to fatigue or frustration | 18 months
  quantitative assessment of the limits of stability in standing done on a force plate (Preuss & Popovic)
Potential for home-based VRT to maintain or improve performance on the Berg Balance Scale | 18 months
  Berg Balance Scale (BBS, Berg et al.)
Potential for home-based VRT to maintain or improve performance on the Timed Up And Go scale (original version) | 18 months
  Timed Up And Go (original version, Campbell et al.)
Potential for home-based VRT to maintain or improve performance on the Timed Up And Go scale (manual version) | 18 months
  Timed Up And Go (manual version, Hofheinz & Schusterschitz)
Potential for home-based VRT to maintain or improve performance on the Timed Up And Go scale (cognitive version) | 18 months
  Timed Up And Go (cognitive version, Lundin-Olsson et al.)
Potential for home-based VRT to maintain or improve performance on the Five Times Sit-To-Stand Test | 18 months
  Five Times Sit-To-Stand Test (FTSST, Bohannon et al.)
Potential for home-based VRT to maintain or improve performance on the Community Balance and Mobility Scale | 18 months
  Community Balance and Mobility Scale (CBM, Howe et al.)
Potential for home-based VRT to maintain or improve performance on quantitative analyses of quiet stance and limits of stability in standing | 18 months
  quantitative analyses of quiet stance and limits of stability in standing (Preuss & Popovic)
Potential for home-based VRT to maintain or improve performance on the Stroke Impact Scale | 18 months
  Stroke Impact Scale (SIS, Duncan et al.)
Potential for home-based VRT to maintain or improve performance on the Reintegration to Normal Living Index | 18 months
  Reintegration to Normal Living Index (RNLI, Spitzer et al).
Determine a sample size for a definitive RCT on home-based VRT | 18 months
  Results of the Berg Balance Scale (BBS, Berg et al.) to calculate sample size.

CONTACTS AND LOCATIONS:
Overall Officials: Hillel Finestone, MD, Principal Investigator — Bruyere Continuing Care
Locations (1):
- Elisabeth Bruyère Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheehy L, Taillon-Hobson A, Sveistrup H, Bilodeau M, Yang C, Welch V, Finestone H. Home-Based Nonimmersive Virtual Reality Training After Discharge From Inpatient or Outpatient Stroke Rehabilitation: Parallel Feasibility Randomized Controlled Trial. JMIR Rehabil Assist Technol. 2025 Mar 28;12:e64729. doi: 10.2196/64729. PMID 40153779
- [Derived] Sheehy L, Taillon-Hobson A, Sveistrup H, Bilodeau M, Yang C, Welch V, Hossain A, Finestone H. Home-based virtual reality training after discharge from hospital-based stroke rehabilitation: a parallel randomized feasibility trial. Trials. 2019 Jun 7;20(1):333. doi: 10.1186/s13063-019-3438-9. PMID 31174579